CLINICAL TRIAL: NCT05778851
Title: Clinical Utility of a Non Endoscopic Device EsoCheck and Biomarker EsoGuard as Alternative to Endoscopy for Screening for Barrett's Esophagus in At Risk Population (ASBE) A Randomized Controlled, Virtual Patient Trial
Brief Title: Clinical Utility of a Non Endoscopic Device EsoCheck and Biomarker EsoGuard as Alternative to Endoscopy for Screening for Barrett's Esophagus in At Risk Population
Acronym: ASBE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lucid Diagnostics, Inc. (Industry)
Collaborators: Medex15 (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Screening
Other Study IDs: ASBE
Record Dates: First submitted 2023-03-10; First posted 2023-03-21 (Actual); Results first posted 2025-10-30 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-03

CONDITIONS: Barrett Esophagus
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Control (No Intervention): Virtual patient cases with GERD and similar BE risk factors as the cases in intervention but without an EsoGuard result and in a different order.
- Intervention (Active Comparator): Virtual patient cases with GERD and similar BE risk factors as the cases in the control arm with an EsoGuard result.
  Interventions: Device: EsoGuard result

INTERVENTIONS:
Device: EsoGuard result — Education slide-set EsoGuard and patient cases including EsoGuard result
  Arms: Intervention

SUMMARY:
This will be a prospective randomized, controlled, virtual, patient study to measure the impact of EsoCheck/EsoGuard on health care provider's decision for upper endoscopy referral.

The participants will complete two rounds of questions concerning the assessed risk for BE and decision for endoscopy referral of 6 patient cases (clinical vignettes).

After the first round has been completed, an EsoCheck/EsoGuard educational information package and the second round of 6 clinical vignettes including EsoGuard results will be sent.

DETAILED DESCRIPTION:
This will be a prospective randomized, controlled, virtual, patient study to measure the impact of EsoCheck/EsoGuard on health care provider's decision for upper endoscopy referral.

Around 200 US physicians will be asked to participate in this study and at least 100 will be enrolled. Physicians eligible for participation are those whose scope of practice includes preventative care and disease screening - namely screening of BE, such as primary care physicians, family medicine physicians, and general practitioners; physicians whose scope of practice include diagnosis and management of esophageal disease may also participate.

The participants will complete two rounds of questions concerning the assessed risk for BE and decision for endoscopy referral of 6 patient cases (clinical vignettes). Per round, there will be 3 different questionnaires consisting of 6 clinical vignettes (A/B/C). Participants will be randomized to questionnaire A, B or C according to the randomization scheme. After the first round has been completed, an EsoCheck/EsoGuard educational information package and the second round of 6 clinical vignettes including EsoGuard results will be sent.

ELIGIBILITY:
Inclusion Criteria:

1. Board-certified physicians whose scope of practice includes preventative care and disease screening, and/or those whose scope of practice include diagnosis and management of esophageal disease (examples include but are not limited to primary care physicians/ general practitioners, family medicine physicians, gastroenterologists, and foregut surgeons);
2. Have between 1 to 40 years of post-residency clinical experience within their field of practice;
3. Have an active panel (whether as part of a group practice, or individually) of over 1000 patients with an adult patient load of more than 50%.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-08-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Victoria T Lee, MD, Principal Investigator — Lucid Diagnostics
Locations (1):
- Lucid Diagnostics, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 97 physicians (participant providers) signed an ICF.
Pre-assignment Details: A total of 90 providers completed the control round questionnaire with 6 control cases (total of 540 control cases) and a total of 87 completed the intervention round questionnaire with 6 cases (total of 522 intervention cases).
Units Other Than Participants: Cases
Groups:
- Participating Physicians: Each participating physician completed 2 times a questionnaire with 6 virtual patient cases per provider with GERD, BE risk factors and without an EsoGuard result and with an EsoGuard result. With 90 participants the total in the control group is 540 control cases, and 87 participants completed the second questionnaire leading to 522 intervention cases.
Period: Overall Study
Arm/Group | Participating Physicians
Started | 90; 540 Cases
Completed | 87; 522 Cases
Not Completed | 3; 18 Cases

BASELINE CHARACTERISTICS:
Groups:
- Participating Physicians: Participating physicians could be primary care physicians or specialists.
Arm/Group | Participating Physicians
Number analyzed (Participants) | 90
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 90
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Data not collected
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Physician type [Count of Participants; unit: Participants] — Population: Primary Care
  Participants
    Primary Care | 68
    Specialist | 22

OUTCOME MEASURES:

1. Primary Outcome: The Impact of EsoCheck/EsoGuard on Provider's Decision for Upper Endoscopy Referral
Description: The change in the percentage/rate of intervention cases who will be referred for endoscopy compared to the control cases.
Time Frame: 1 month
Population: A total of 540 control cases were reviewed by 90 providers, and a total of 522 intervention cases were reviewed by 87 providers.
Measure: Number; unit: Cases
Units Other Than Participants: Cases
Groups:
- Control Cases: Virtual patient cases without EsoGuard results
- Intervention Cases: Virtual patient cases with EsoGuard results
Arm/Group | Control Cases | Intervention Cases
Number analyzed (Participants) | 90 | 87
Number analyzed (Cases) | 540 | 522
Cases | 382 | 211

2. Secondary Outcome: The Impact of EsoCheck/EsoGuard on Provider's Decision for Upper Endoscopy Referral for EsoGuard Positive Cases
Description: The change in the percentage/rate of EsoGuard postive intervention cases who will be referred for endoscopy compared to the control cases.
Time Frame: 1 month
Population: A total of 90 EsoGuard + control cases were reviewed by 90 providers, and a total of 87 EsoGuard + intervention cases were reviewed by 87 providers.
Measure: Number; unit: Cases
Units Other Than Participants: Cases
Arm/Group | Control Cases | Intervention Cases
Number analyzed (Participants) | 90 | 87
Number analyzed (Cases) | 90 | 87
Cases | 53 | 78

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Groups:
- Participants: Physician providers who completed online questionnaires
Arm/Group | Participants
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-06): https://cdn.clinicaltrials.gov/large-docs/51/NCT05778851/Prot_SAP_001.pdf